CLINICAL TRIAL: NCT03333967
Title: The Real World Study of Apatinib for Gastric Cancer Treatment in Anhui Province
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: AHAT-104
Record Dates: First submitted 2017-10-01; First posted 2017-11-07 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-09

CONDITIONS: Gastric Cancer
Keywords: apatinib
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators conduct the real world study to explore the efficacy and safety of Apatinib in gastric cancer .

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients .
2. Confirmed by Pathology or histology of Gastric cancer
3. Patients should be voluntary to the trial and provide with signed informed consent
4. The researchers believe patients can benefit from the study.

Exclusion Criteria:

1. Patients with a known history of allergic reactions and/or hypersensitivity attributed to apatinib or its accessories
2. Pregnant or lactating women
3. Patients with Apatinib contraindications
4. Patients of doctors considered unsuitable for the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients of gastric cancer in Anhui province
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-09-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Progress free survival | 1 year
  Progress free survival is defined as the length of time from random assignment to disease progression or to death resulting from any cause other than the progress.

SECONDARY OUTCOMES:
disease control rate | 1year
  Investigators will assess treatment response according to Response Evaluation Criteria in Solid Tumors 1.1
Objective tumor response rate | 1year
  Objective tumor response rate is defined as the percentage of subjects having achieved confirmed Complete Response + Partial Response as best overall response according to radiological assessments
overall survival | 3year
  overall survival is defined as the length of time from random assignment to death or to last contact.
Disease-free survival | 1 year
  Disease-free survival is defined as the length of time from the date of randomization to the date of first documentation of relapse of gastric cancer or any other type of cancer or death.

OTHER OUTCOMES:
Quality of life score | 1year
  Quality of life score is a questionnaire developed to assess the quality of life of cancer patients.
adverse events | 1year
  adverse events are evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events v4.0.

CONTACTS AND LOCATIONS:
Overall Officials: China Anhui, Study Chair — The First Affiliated Hospital of Anhui Medical University
Locations (1):
- First Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Peng W, Zhang F, Wang Z, Li D, He Y, Ning Z, Sheng L, Wang J, Xia X, Yu C, Wang Z, Zhao Y, Liang H, Hu B, Sun C, Wang D, Cheng Y, Pan M, Xia L, Guo X, Zhang Y, Hu Z, Li X, Lu L, Zhang J, Qian H, Xie H, Sun G. Large Scale, Multicenter, Prospective Study of Apatinib in Advanced Gastric Cancer: A Real-World Study from China. Cancer Manag Res. 2020 Aug 6;12:6977-6985. doi: 10.2147/CMAR.S249153. eCollection 2020. PMID 32821164
- [Derived] Du Y, Cao Q, Jiang C, Liang H, Ning Z, Ji C, Wang J, Zhou C, Jiang Z, Yu C, Li L, Zhao Y, Xu Y, Xu T, Hu W, Wang D, Cheng H, Wang G, Zhou J, Wang S, Zhang Y, Hu Z, Li X, Lu D, Zhang J, Xie H, Sun G. Effectiveness and safety of low-dose apatinib in advanced gastric cancer: A real-world study. Cancer Med. 2020 Jul;9(14):5008-5014. doi: 10.1002/cam4.3105. Epub 2020 May 22. PMID 32441892